CLINICAL TRIAL: NCT01257646
Title: Observation of the Gait Cycle in Patients With Hemiplegia in Order to Improve the Triggering of Functional Electrical Stimulation
Acronym: MASEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LOCAL/2009/JF-01; 2010-A00534-35 (Other: RCB number)
Record Dates: First submitted 2010-12-09; First posted 2010-12-10 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2015-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Gait Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Recent stroke group (Experimental): These patients have hemiplegia following a stroke within the last 6 months
  Interventions: Other: Gait analysis
- Old stroke group (Active Comparator): The patients have hemiplegia following a stroke that took place at least a year ago
  Interventions: Other: Gait analysis

INTERVENTIONS:
Other: Gait analysis — A Gaitrite system, a goniometer, and EMG are used to record data while the patient walks 10 meters.

SUMMARY:
The main objective of this study is the estimation and comparison of the dephasing between the switch heel and the inertial placed on the paretic foot compared to the events of the gait cycle determined by a Gaitrite system (beginning and end of the swing phase) in conditions without stimulation.

ELIGIBILITY:
Inclusion Criteria:

* patient has had a first ischemic or hemorragic stroke (supratentorial) within the last 6 months for the "recent stroke" group, or more than a year ago for the "old stroke" group
* the patient can walk 10 m without human help, with or without a cane, and a deficit of the foot levator requiring the use of technical assistance to remedy this or involving walking problems
* electrostimulated contraction of the anterior tibialis is possible
* patient has been informed and has signed the consent form

Exclusion Criteria:

* cognitive disorder making participation in the study difficult
* fixed plantar flexion, knee extended below 0°
* patient refuses to sign consent
* patient is not covered by a social security system
* patient is under any kind of guardianship

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Timing of heel strike (s) | 10 seconds
  The goal is to use the data generated by this observational study to predict the timing of the heel strike when a patient walks.

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme Froger, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- Centre Hospitalier Universitaire de Nîmes, Nîmes, Gard, France